CLINICAL TRIAL: NCT02261350
Title: The Effect of Nutritional Support on Gait Speed Following Hospitalisation for Acute Exacerbation of COPD
Brief Title: Post-hospitalisation Nutritional Support and Gait Speed in COPD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Medical Research Council (Other Government); The Hillingdon Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2013LF004H
Record Dates: First submitted 2014-05-08; First posted 2014-10-10 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Respiratory Tract Diseases; Lung Diseases, Obstructive; Bronchitis, Chronic; Pulmonary Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Tract Diseases; Lung Diseases, Obstructive; Bronchitis, Chronic; Pulmonary Emphysema | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Food Fortification (Experimental): Food Fortification
  Interventions: Dietary Supplement: Food fortification
- Oral Nutritional Supplements (Experimental): Oral Nutritional Supplements - Fortisip Compact
  Interventions: Dietary Supplement: Oral Nutritional Supplements
- Usual Care (No Intervention)

INTERVENTIONS:
Dietary Supplement: Food fortification
  Arms: Food Fortification
Dietary Supplement: Oral Nutritional Supplements
  Other Names: Fortisip Compact, Nutricia Clinical
  Arms: Oral Nutritional Supplements

SUMMARY:
To determine the feasibility of delivering different community nutritional interventions to chronic obstructive pulmonary disease (COPD) patients at moderate or severe risk of malnutrition following a hospitalisation for an acute exacerbation of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Ability to consent
* Patients at moderate or severe risk of malnutrition
* Adults over the age of 40
* Hospitalised with an AECOPD

Exclusion Criteria:

* Receiving long term parental or enteral nutrition
* Inability to swallow or difficulty liquids
* Lactose intolerance, galactosaemia, cow's milk protein allergy or intolerance
* Co-existing active cancer, progressive neurological condition or active GI disorder.
* Receiving palliative care with expectation of death within 3 months
* Cognitive dysfunction or unable to consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in four-metre gait speed (m/s) following nutritional support | Change from baseline to 12 weeks

SECONDARY OUTCOMES:
Change in weight (kg) following nutritional support | Change from baseline to 12 weeks
Change in fat free mass (kg) as measured by bioelectrical impedence following nutritional support | Change from baseline to 12 weeks
Change in fat free mass index (kg/m2) as measured by bioelectrical impedence following nutritional support | Change from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Man, PhD FRCP, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- The Hillingdon Hospital NHS Foundation Trust, Uxbridge, Middlesex, United Kingdom